CLINICAL TRIAL: NCT00803036
Title: Spreading Depressions as Secondary Insults After Traumatic Injury to the Human Brain
Brief Title: Observational Study of Cortical Spreading Depression in Human Brain Trauma
Acronym: COSBID-TBI
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: University of Miami (Other); University of Pittsburgh (Other); Virginia Commonwealth University (Other); King's College London (Other)
Responsible Party: Principal Investigator, Jed Hartings, Associate Research Professor, University of Cincinnati
Other Study IDs: 08-96-12-01; CDMRP-W81XWH-08-2-0016
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Traumatic Brain Injury
Keywords: spreading cortical depression; electroencephalography; traumatic brain injury; intensive care; vascular hypotension; intracranial hypertension
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypotension; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Since the primary damage from traumatic brain injury (TBI) is irreversible, the focus of medical management of TBI is preventing secondary injury that can be life-threatening and worsen patient outcome. Insight into the pathologic mechanisms of secondary injury, which are largely unknown, is required for developing better treatments.

In preliminary studies, the investigators have found that a pathologic brain activity, known as spreading depression, recurs in a large number of TBI patients in the first week after injury. Spreading depressions are short-circuits of brain function that arise spontaneously from an injury and spread repeatedly as waves into neighboring brain tissue. Animal research has shown that spreading depressions can cause secondary injury to the brain.

The primary objective of this observational study is to determine whether the occurrence or severity of spreading depression is related to worse neurologic recovery from TBI. Results from the study will determine whether monitoring of spreading depression should be used as a guide or target for improved medical management of the TBI patient.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* diagnosis of TBI
* craniotomy performed as per required treatment of TBI
* craniotomy surgery < 7 days after TBI
* GCS<13 at time of decision for surgery
* expected neuromonitoring for >72 hr

Exclusion Criteria:

* any failure to meet above criteria
* pregnancy
* GCS 3 with fixed, dilated pupils

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to study hospitals who require neurosurgery for acute traumatic brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incidence of spreading depressions as assessed by continuous electrocorticography for 3-7 days after surgery. Primary neurologic outcome will be measured by the Glasgow Outcome Score - Extended. | Six months post-TBI.

SECONDARY OUTCOMES:
Post-traumatic epilepsy questionnaire. | 6, 12, and 24 months post-TBI

CONTACTS AND LOCATIONS:
Overall Officials: Jed A. Hartings, PhD, Principal Investigator — University of Cincinnati
Locations (5):
- United States (4):
  - University of Miami, Miami, Florida
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
- King's College Hospital, London, United Kingdom

REFERENCES:
- See also: This study is conducted as a branch of COSBID, the Co-Operative Study of Brain Injury Depolarizations. — http://www.cosbid.org